CLINICAL TRIAL: NCT02816528
Title: Efficacy of Information System Regarding the Consumption of Antibiotics and Bacterial Resistance on the Use of Antibiotics in Primary Care
Brief Title: Efficacy of Information System Regarding the Consumption of Antibiotics and Bacterial Resistance in Primary Care
Acronym: SICAR-Amb
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Direction Générale de l'Offre de Soins (Other Government); CNAMTS, Caisse Nationale d'Assurance Maladie des Travailleurs salariés, France (Unknown); MedQual, Nantes, France (Unknown)
Responsible Party: Sponsor
Other Study IDs: PREPS-15-000171
Record Dates: First submitted 2016-06-10; First posted 2016-06-28 (Estimated); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Chronic Disease
Keywords: Antibiotics; Primary care; Stewardship; General practitioners
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Training program: Physicians will be given informations regarding antibiotic consumptions and bacterial resistance in their activity area every 3 months during 12 months.
  Interventions: Behavioral: Training program
- Nothing: Not Trained Physicians

INTERVENTIONS:
Behavioral: Training program — Physicians will be given informations regarding antibiotic consumptions and bacterial resistance in their activity area every 3 months during 12 months.
  Groups: Training program

SUMMARY:
France is a country strong consumer of antibiotics in Europe, specially in primary care.

Outpatient antibiotic use represents around 90% of total antibiotic use and prescriptions come mainly from general practitioners. A literature review of antibiotic stewardship in primary care show that there is no evaluation of interest of giving information about consumption of antibiotics and bacterial resistance to general practitioners. The objective of this study is to demonstrate that practitioners implicated in the followed of consumption of antibiotics and bacterial resistance around their geographical area of practice could change and improve their practices in good use of antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* General practitioners in a "Meurthe-et-Moselle" french department

Exclusion Criteria:

* General practitioners out of "Meurthe-et-Moselle" french department

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: General practitioners
Sampling Method: Non-Probability Sample
Enrollment: 472 (Estimated)
Dates: Start 2016-06-24 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Consumption of antibiotics | 36 months
  Antibiotics consumptions are provided by CNAMTS and calculated in defined daily dose DDD/1000 patient-days around the geographical area concerned by this study.

SECONDARY OUTCOMES:
Bacterial resistance of Escherichia coli and Staphylococcus aureus | 36 months
  The number of intermediate and resistant strains of E.coli and S.aureus are provided by MedQual around the geographical area concerned by this study.

CONTACTS AND LOCATIONS:
Overall Officials: Béatrice DEMORE, Principal Investigator — Centre Hospitalier Régional Universitaire, Brabois, Pharmacy

IPD SHARING:
Plan to Share IPD: Undecided